CLINICAL TRIAL: NCT05125094
Title: Prognostic Performance of Preoperative and Follow up by Gadoxetic Acid-Enhanced MRI in Patients With HCC After TACE Combined With Ablation: Compared With Non-gadoxetic Enhanced MRI
Brief Title: Prognostic Performance of Preoperative and Follow by Gadoxetic Enhanced MRI in HCC Patients After TACE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2020-060R
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma Stage III
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Gadoxetic MRI for diagnosis: the patients with HCC follow up with Non-Gadoxetic MRI for diagnosis
  Interventions: Device: TACE,Ablation
- Gadoxetic MRI for diagnosis: the patients with HCC follow up with Gadoxetic MRI for diagnosis
  Interventions: Device: TACE,Ablation

INTERVENTIONS:
Device: TACE,Ablation — Transcatheter arterial chemoembolization

SUMMARY:
Interventional therapy is an effective alternative for patients with hepatocellular carcinoma (HCC) who are not indicated for surgery. CT or MRI imaging findings are important diagnostic and evaluation criteria for preoperative diagnosis and postoperative efficacy evaluation of TACE. In addition, the recurrence rate of liver cancer is very high, even with radical treatment, the 5-year recurrence rate is still as high as 70%. Therefore, postoperative follow-up and early detection of recurrent lesions by imaging are beneficial to the prognosis and survival benefit. Gadoxetic acid is a liver-specific MRI contrast agent for the diagnosis of liver cancer, especially in early stage, or small liver cancer (<2cm). Therefore, gadoxetic acid enhanced MRI is very important for the decision making and prognosis of HCC patients. TACE combined with ablative therapy has received clinical attention, which can significantly improve the clinical efficacy and reduce liver function damage. The study forces on evaluating the changes in survival in patients with liver cancer who were scheduled to receive TACE combined with ablation and regularly followed up, compared with enhanced CT or conventional MRI as imaging assessment (preoperative diagnosis and postoperative follow-up).

DETAILED DESCRIPTION:
China is a country with a high incidence of hepatocellular carcinoma (HCC), and the number of new cases of HCC every year accounts for more than 50% of the world, while the diagnosis rate of very early and early HCC patients in China only accounts for about 25%, and most patients cannot be operated on. Interventional therapy is an effective alternative for patients with hepatocellular carcinoma (HCC) who are not indicated for surgery. CT or MRI imaging findings are important diagnostic and evaluation criteria for preoperative diagnosis and postoperative efficacy evaluation of TACE. In addition, the recurrence rate of liver cancer is very high, even with radical treatment, the 5-year recurrence rate is still as high as 70%. Therefore, postoperative follow-up and early detection of recurrent lesions by imaging are beneficial to the prognosis and survival benefit. Currently, the main clinical follow-up methods are enhanced CT and non-gadoxetic acid enhanced magnetic resonance examination. Gadoxetic acid is a liver-specific MRI contrast agent for the diagnosis of liver cancer, especially in early stage, or small liver cancer (<2cm). Compared with enhanced CT alone, the combination of Gadoxetic acid MRI for pre-treatment diagnosis of early-stage HCC significantly improved 4-year survival. Therefore, gadoxetic acid enhanced MRI is very important for the decision making and prognosis of HCC patients. TACE combined with ablative therapy has received clinical attention, which can significantly improve the clinical efficacy and reduce liver function damage. Currently, there are few studies on the survival rate of liver cancer patients receiving TACE combined with ablative therapy with gadoxetic acid enhanced MRI. The study forces on evaluating the changes in survival in patients with liver cancer who were scheduled to receive TACE combined with ablation and regularly followed up, compared with enhanced CT or conventional MRI as imaging assessment (preoperative diagnosis and postoperative follow-up).

ELIGIBILITY:
Inclusion Criteria:

Patients who will be initially diagnosed as HCC and plan to receive TACE, or combined with ablation as first-line treatment Age from 18 - 75 Sign ICF （Informed consent form） mainly stage B patients with Child-Pugh class A or B liver function and an ECOG score of 0-2; multiple nodular tumors; a main portal vein that is not completely blocked or is completely blocked but the compensatory collateral blood vessels have formed between the hepatic artery and portal vein

Exclusion Criteria:

Women who are pregnant, lactating Contraindications to MRI Contrast media: Hypersensitivity General contraindications to MRI such as pacemaker, severe claustrophobia etc. Patients who received or plan to take other treatment (resection, chemical, immunotherapy drugs that will systemic effect survival) before TACE combined with ablation

Patients with Contraindications of TACE or ablation :

1. Severe liver dysfunction (Child-Pugh class C), including jaundice, hepatic encephalopathy, refractory ascites, or hepatorenal syndrome;
2. severe coagulation dysfunction that cannot be corrected;
3. completely embolized main portal vein with few collateral blood vessels formed;
4. wide distant metastasis with an estimated survival of < 3 months;
5. significant reductions in peripheral blood leukocytes and platelets, white blood cell (WBC) count < 3.0 × 109/L (when due to hypersplenism but not toxicity of chemotherapy; therefore, it is not an absolute contraindication for TACE), and platelets < 50 × 109/L;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are initially diagnosed as HCC will plans to receive first curative TACE combined with ablation and can be followed up in the hospital with contrast enhanced MRI
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | mean follow up 34 months
  Comparison of Overall Survival after TACE combined with ablation between the Two Groups

SECONDARY OUTCOMES:
tumor response | mean follow up 34 months
  Comparison of tumor response after TACE combined with ablation between the Two Groups

CONTACTS AND LOCATIONS:
Overall Officials: Mengsu Zeng, PhD, Study Director — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: No
The results of this study may be published in medical journals, but we will keep patient information confidential as required by law, and patient personal information will not be disclosed unless required by relevant law.

REFERENCES:
- [Result] Guo J, Seo Y, Ren S, Hong S, Lee D, Kim S, Jiang Y. Diagnostic performance of contrast-enhanced multidetector computed tomography and gadoxetic acid disodium-enhanced magnetic resonance imaging in detecting hepatocellular carcinoma: direct comparison and a meta-analysis. Abdom Radiol (NY). 2016 Oct;41(10):1960-72. doi: 10.1007/s00261-016-0807-7. PMID 27318936
- [Result] Lan H, Lin G, Zhong W. A meta-analysis of the added value of diffusion weighted imaging in combination with contrast-enhanced magnetic resonance imaging for the diagnosis of small hepatocellular carcinoma lesser or equal to 2 cm. Oncol Lett. 2020 Sep;20(3):2739-2748. doi: 10.3892/ol.2020.11805. Epub 2020 Jul 3. PMID 32782590